CLINICAL TRIAL: NCT04663503
Title: Benefits of Intrahospital Exercise Program in Pediatric Hematopoietic Stem Cell Transplant-A Randomized Control Trial
Brief Title: Benefits of Exercise Program in Pediatric HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Alex Ngwube, Assistant Professor, Phoenix Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-16-127
Record Dates: First submitted 2020-08-26; First posted 2020-12-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Exercise; Transplantation
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm -Exercise Program (Experimental): This structured exercise program will incorporate a specially designed, low intensity, resistance based exercise regime created by our physical therapist. It consists of strengthening, endurance, stretching and relaxation exercises tailored according to age and their ability to perform activities throughout their hospitalization (Appendix 3). This exercise program will be done three times a week for 30-45 mins supervised by the same physiotherapist throughout hospitalization and will be self-administered every weekend. A home exercise program printout with the appropriate resistance exercises will be provided to the family upon discharge, with instructions on how often to complete throughout the week. Discharged children will attend one supervised exercise session per week with the physiotherapist for six weeks. The family and patient will also be provided a weekly sheet to check off the days they completed strengthening and endurance exercises.
  Interventions: Other: Exercise program
- Control arm- No intervention (No Intervention): The second arm of the study involves patients following standard of care during the HSCT period in the hospital with PT evaluation and management prescribed as needed by their transplant medical team including any additional PT interventions as a result of clinical indications. No additional intervention is incorporated in this group

INTERVENTIONS:
Other: Exercise program — Depending on the age, there will be two components of the exercise program completed by the patients. The first component will be strengthening exercises. The second component will be endurance activities. This will be administered by the physical therapist
  Arms: Intervention arm -Exercise Program

SUMMARY:
Deconditioning is a common adverse effect of short and long-term immobilization. For months pediatric hematopoietic stem cell transplant patients can be quarantined while hospitalized, much of which time is spent immobilized putting these patients at a higher risk for loss of muscle strength, functionality, endurance, and quality of life. Phoenix Children's Hospital is conducting approximately forty (40) transplants per year. Adult studies have shown that exercise as an effective counter measure to deconditioning in stem cell transplant patients. However, there is a knowledge gap in pediatric HSCT. Thus this study is being conducted to determine if there is a correlation between intra-hospital exercise and improved functionality, mobility, strength, and quality of life. To achieve these aims investigators will perform a randomized control study. The investigators will aim to recruit 40 patients, 20 in each arm, ages 4-21 at Phoenix Children's Hospital. Each participant will receive baseline measures by a physical therapist; for functionality using (WeeFIM), muscle strength using manual muscle testing (MMT), endurance using the 6-minute walk test, and quality of life using the NIH PROMIS measures. Measurements will be taken again at discharge and 6-weeks post-discharge. During hospital admittance the intervention group will perform exercise routines 3 times weekly while the control group will be treated per standard of care with no exercise intervention. Patients recruited must be receiving first HSCT. A full explanation of the study and possible benefits will be given to the patients and their families upon consent. Primary outcomes will look at endurance, functionality and muscle strength. Secondary outcomes will include QoL and amount of achievable "time out of bed".

DETAILED DESCRIPTION:
Despite growing numbers of publications describing the effects of these exercise modalities in adult HSCT patients, only limited attention has been paid to this effective supportive therapy in children. Only five publications describe the effectiveness of exercise training in pediatric HSCT. San Juan et al. showed beneficial effects on functional performance, muscle strength, and Qol scores in a study of children (aged 8-16) undergoing a supervised exercise program that included resistance and aerobic exercises for 3 weeks after HSCT. In another study, the moderate intensity exercise program implemented to children undergoing allogeneic HSCT for 3 weeks during hospitalization showed positive effects on body mass and body mass index (BMI), and no negative effect on immune cell recovery. It was found that a structured physical activity program has positive effects on Qol and fatigue scores in children undergoing peripheral blood stem cell transplantation. Yildez et al. showed improvement in areas such as functional performance, muscle strength, functional mobility. Marchese et al. showed an improvement in knee extension strength and ankle dorsiflexion range of motion.This study will implement an exercise program that is personalized to hematopoietic stem cell transplant recipients designed to prevent a decline in function/independence. Investigators will accomplish this by conducting a randomized controlled trial (RCT) that will examine the effect of an 8-12 week personalized exercise program compared to standard care following hematopoietic stem cell transplantation. Data from this study should increase understanding of the effect of exercise in this population on QoL, functional ability, endurance, muscle strength, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 4-21 years
* Admitted for Hematopoietic Stem Cell Transplant

Exclusion Criteria:

* Patients with any preexisting need for gait assistance such as crutches, wheelchair, braces, or walker
* Previous Stem Cell Transplant in the last 6 months
* Patients with grade 3 or greater sensory/motor neuropathy

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | Change from baseline at enrollment, to discharge from hospital and at 6 weeks post discharge
  Used in measuring exercise capacity and endurance.
Pediatric Functional Independence Measure (WeeFIM) | Change from baseline at enrollment, to discharge from hospital and at 6 weeks post discharge. This would be done through study completion, an average of 12 weeks.
  Used to measure functionality.
Manual muscle testing (MMT) | Change from baseline at enrollment, to discharge from hospital and at 6 weeks post discharge.This would be done through study completion, an average of 12 weeks.
  Useful to measure muscle strength

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Measures | Change from baseline at enrollment, to discharge from hospital and at 6 weeks post discharge. This would be done through study completion, an average of 12 weeks.
  Changes in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ngwube, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith C, Farhat R, Fern-Buneo A, Purrington H, Cobb E, Matson L, Kang P, Beebe K, Campbell C, Schwalbach C, Salzberg D, Miller H, Adams R, Ngwube A. Effects of an exercise program during pediatric stem cell transplantation: A randomized controlled trial. Pediatr Blood Cancer. 2022 May;69(5):e29618. doi: 10.1002/pbc.29618. Epub 2022 Feb 23. PMID 35195344